CLINICAL TRIAL: NCT01282983
Title: Study of Digestive Tolerance of Orange Juice With Fibers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Dan Linetzky Waitzberg - Professor, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IKEA2010
Record Dates: First submitted 2011-01-20; First posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-10

CONDITIONS: Digestive Alteration [PE]
Keywords: fiber; orange juice; digestive symptom
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fiber (Active Comparator)
  Interventions: Dietary Supplement: Fiber
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fiber — The study consists of 21 days consumption of Orange juice. The volunteers will be instructed to consume 200ml of juice twice a day (1 pack of 200ml at lunch and one at dinner) with 4grams of fiber in each pack.
  Arms: fiber
Dietary Supplement: Placebo — The study consists of 21 days consumption of Orange juice. The volunteers will be instructed to consume 200ml of juice twice a day (1 pack of 200ml at lunch and one at dinner) without fiber.
  Arms: Placebo

SUMMARY:
Dietary fiber (commonly called bulk or roughage) is the edible nondigestible component of carbohydrate and lignin naturally found in plant food; however, bacteria in the lower gut may metabolize part of it. Epidemiological studies have found that fiber intake in the population is below the suggested recommendations. The beneficial effects of the fibers in human health are recognized. The regular intake of dietary fiber has an important role in the intestinal function increasing the intestinal fecal and reducing the transit time along the intestine; collaborates with the LDL-cholesterol plasmatic reduction by increasing fecal excretion of cholesterol and bile acids, decreases postprandial glucose in healthy, diabetics and insulin resistant people, reduces the risk for developing certain cancers, promotes satiety, helps with weight loss, and exerts immunomodulatory effect. However, fiber intake may be associated with adverse effects such as flatulence, bloating, cramps, and daily consumption of orange juice to bring digestive problems associated with acidity and heartburn, epigastric burning. Then it becomes of interest to study the tolerance of a new orange juice product fortified with mixed fibers (fructooligosaccharides, resistant dextrin, polydextrose and lactulose).

DETAILED DESCRIPTION:
Monocentric, double blind, randomized, two parallel arms controlled placebo study. 200 healthy women from 18 to 45 years old, without functional digestive disorders or diagnosed digestive disease will take part in the study. The study consists of 21 days consumption of Orange juice. The participants will be randomized in two groups: placebo (Orange juice without fiber - control) and study group (Orange juice fortified with fiber mix). In both groups, the volunteers will be instructed to consume 200ml of juice twice a day (1 pack of 200ml at lunch and one at dinner).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Tolerate the intake of orange juice routinely (at least twice/month)
* Do not use antibiotics, industrial fibers or supplements containing industrialized fibers, prebiotics and probiotics for 30 days before the start of the study
* BMI between 18,5 a 29,9 Kg/m2
* Body weight stable during the last two months
* Able to have good communication with the researcher
* Understand and agree with the rules of the study
* Making use of some contraceptive method
* Non-smokers (less than five cigarettes/day)

Exclusion Criteria:

* Illiterate
* Severe alcoholics
* Allergy to orange and its juice
* Any other allergy or food intolerance
* Disease or disorder of the upper digestive tract diagnosed and treated in the last twelve months
* Inflammatory bowel diseases
* Irritable bowel syndrome
* To have diarrhea (three liquid evacuations a day)
* Pregnancy
* Lactation
* Any history of eating disorder
* Declared diseases:

  * Renal insufficiency
  * Hepatic Insufficiency
  * Chronic Heart Failure
  * Other disease which in the opinion of the investigator might be inconsistent with the study
* Be in dialysis process
* Chronic renal failure
* History or evidence of organic disease of the gastrointestinal tract
* History of cancer within five previous years (except basal cell carcinoma well treated or cervical carcinoma in situ)
* History or evidence of metabolic disturbs
* History of gastric surgery intervention (except appendectomy)
* Being under some weight loosing process or diet
* Refuse to sign the Informed Consent Term

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-02 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of stool - Chart | Frequency of stool - Chart
  Bristol scale with classification type 1 to type 7 will be used for self-information on daily frequency of bowel movements and consistency of the feces.

SECONDARY OUTCOMES:
Unwanted symptoms classification | Unwanted symptoms classification
  The daily graduation of nuisance for abdominal pain, flatulence, abdominal distension, nausea and vomiting using the classification for unwanted symptoms, with 4-point scale, after 3 weeks consumption of product with the information obtained with the standard orange juice consumption from the participant diary

CONTACTS AND LOCATIONS:
Overall Officials: Dan L Waitzberg, MD PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil